CLINICAL TRIAL: NCT02620462
Title: Explore the Effectiveness of a Sensor-based Interactive Exercise Training on Functional Performance in Patients With Knee Osteoarthritis
Brief Title: Wearable Sensor-based Balance Training for Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Bijan Najafi, Associate Prof, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1501657972
Record Dates: First submitted 2015-06-08; First posted 2015-12-03 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Knee Osteoarthritis
Keywords: Postural Balance; Pain; Gait; Physical Activity Level
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wearable sensor-based exercise training (Experimental): The intervention group in addition to standard of care, will receive 6 weeks of sensor-based balance training that provides real-time visual feedback of lower extremities during exercise. The visual feedback is provided on computer screen.
  Interventions: Device: Wearable sensor-based exercise training
- Control Group (No Intervention): The control group only receives standard of care.

INTERVENTIONS:
Device: Wearable sensor-based exercise training — The device provides real-time visual feedback of joint movement during balance exercise
  Arms: Wearable sensor-based exercise training

SUMMARY:
Knee osteoarthritis (KOA) is one of the leading causes of lower limb disability among the elderly and can cause loss of knee joint proprioception that contributes towards deterioration of postural balance. Maintaining a good postural stability is essential while performing everyday functional activities and to avoid falls. Exercise training has been reported to reduce pain as well as improve performance of functional tasks in patients with KOA however compliance to exercise can be challenging due to pain, lack of motivation and traditional nature of exercise that can easily overtax patients. Furthermore, there are not exercise programs that are specifically designed for patients with KOA in order to address lost knee joint proprioception. Recent studies have also demonstrated that visual feedback during exercise can enhance the benefits of exercise training. Therefore, the aim of the proposed study is to implement an interactive sensor-based exercise training to improve postural balance, gait and activities of daily living in patients with KOA.

DETAILED DESCRIPTION:
The exercise intervention procedure is based on wearable sensor game-based balance-training program (Exergame). Subjects will perform progressive balance exercises such as ankle reaching or weight shifting, obstacle crossing, and ankle trail making task (i.e. motor-cognitive task). Real-time visual/audio lower-extremity joint motion feedback will be provided using wearable sensors (LEGSys, Biosensics LLC, Cambridge, MA, USA) to assist and encourage subjects to accurately execute each exercise task. The same wearable sensor technology is also used to quantify changes in balance and gait.

Changes in balance, gait, fear of falling, physical activity, pain, and quality of life parameters will be assessed at the beginning and conclusion of the training program.

Subjects will perform sensor-based interactive balance training (on computer screen), 2 x week, for a period of 6 weeks. The training consists of three balance tasks shown on a computer screen (1. ankle reaching task or weight shifting , 2. obstacle negotiation task, and 3. ankle trail making task (i.e. motor-cognitive task) intended to improve postural stability.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above
* ability to walk 50 m independently (with or without aid)
* ability to stand for 5 minutes .

Exclusion Criteria:

* disorder other than osteoarthritis that may severely affect gait and balance

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Body Sway as an indicator of postural control | 6 weeks
  Body sway including ankle sway, hip sway, and center of mass sway

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | 6 weeks
  Knee injury and Osteoarthritis Outcome Score measured by KOOS
Gait | 6 weeks
  Spatio-temporal parameters of gait including gait speed, double support, and stride length
Pain | 6 weeks
  Pain intensity will be assessed using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Bijan Najafi, PhD, Principal Investigator — University of Arizona
Locations (1):
- The University of Arizona Arthritis Center, Tucson, Arizona, United States